CLINICAL TRIAL: NCT02658461
Title: Time and Motion Study of Trastuzumab Subcutaneous (SC) and Intravenous (IV) Formulations for the Treatment of Patients With HER2-Positive Early Breast Cancer (EBC)
Brief Title: An Observational Time and Motion Study of Trastuzumab Subcutaneous (SC) and Intravenous (IV) Formulations in Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Early Breast Cancer (EBC)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29123; 2010-024099-25 (EudraCT Number)
Record Dates: First submitted 2016-01-11; First posted 2016-01-18 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Trastuzumab IV Infusion: Participants with HER2-positive EBC will be evaluated for the costs and other factors associated with health care utilization with the administration of trastuzumab via IV infusion.
  Interventions: Drug: Trastuzumab
- Trastuzumab SC Single-Use Injection Device: Participants with HER2-positive EBC will be evaluated for the costs and other factors associated with health care utilization with the administration of trastuzumab via SC single-use injection device.
  Interventions: Drug: Trastuzumab
- Trastuzumab SC Vial/Syringe: Participants with HER2-positive EBC will be evaluated for the costs and other factors associated with health care utilization with the administration of trastuzumab via SC vial/syringe.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab will be given on Day 1 of each 3-week cycle for a total of 18 cycles. Dosage will be according to the local labeling: 600 milligrams (mg) SC or 6 milligrams per kilogram (mg/kg) via IV infusion. For those assigned to the IV arm or if IV treatment is delayed >1 week, an initial loading/reloading dose of 8 mg/kg will be given instead. Due to the observational nature of this study, trastuzumab is not an investigational product but will be supplied in the MO22982 trial. Each route/device (SC single-use injection device, SC vial/syringe, IV infusion) will be observed in at least 12 episodes of care.
  Other Names: Herceptin

SUMMARY:
This prospective, non-interventional time and motion study will evaluate the costs of healthcare resource utilization associated with the administration of trastuzumab (Herceptin) SC and IV formulations in HER2-positive EBC. This is a sub-study of the clinical study MO22982 (NCT01401166/PrefHer).

ELIGIBILITY:
Inclusion Criteria:

* Participants from the MO22982 (PrefHer) clinical trial who consent to the presence of an observer to record data for the study during administration of trastuzumab
* Members of the care team responsible for management of participants from the MO22982 (PrefHer) clinical trial who also consent to the presence of an observer during administration of trastuzumab

Exclusion Criteria:

* None specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult females with HER2-positive EBC who participated in the parent study MO22982 will be observed in this non-interventional study.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United Kingdom (4):
  - Brighton
  - Cardiff
  - Maidstone
  - Nottingham

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants from the MO22982 (NCT01401166) trial were observed for this time and motion study of trastuzumab. The focus of the observation in this study was the HCP rather than the person being treated, so number of observations is reported everywhere instead of number of participants. Number of participants was not collected.
Pre-assignment Details: Each arm included 12 observations of an episode of care independent of the person being treated. By design of the study, some individuals may have been observed more than once and there may have been fewer than 12 actual participants in each arm. As only a single observation was required to participate, there was no "disposition" recorded.
Groups:
- Trastuzumab Single-Use Injection Device: Participants with human epidermal growth factor receptor 2 (HER2)-positive early breast cancer (EBC) received trastuzumab via single-use injection device as 600 milligrams (mg) on Day 1 of each 3-week cycle for a total of 18 cycles. Trastuzumab was supplied in the MO22982 (NCT01401166) trial and dosed according to local labeling.
- Trastuzumab Subcutaneous (SC) Injection: Participants with HER2-positive EBC received trastuzumab via SC injection using vial/syringe as 600 mg on Day 1 of each 3-week cycle for a total of 18 cycles. Trastuzumab was supplied in the MO22982 (NCT01401166) trial and dosed according to local labeling.
- Trastuzumab Intravenous (IV) Infusion: Participants with HER2-positive EBC received trastuzumab via IV infusion as 6 milligrams per kilogram (mg/kg) on Day 1 of each 3-week cycle for a total of 18 cycles. An initial loading dose of 8 mg/kg was given during the first cycle, and also reserved as a reloading dose if treatment was delayed greater than (>) 1 week. Trastuzumab was supplied in the MO22982 (NCT01401166) trial and dosed according to local labeling.
Period: Overall Study
Arm/Group | Trastuzumab Single-Use Injection Device | Trastuzumab Subcutaneous (SC) Injection | Trastuzumab Intravenous (IV) Infusion
Started | 12 (The enrollment reflects episodes of care and not number of actual participants.) | 12 (The enrollment reflects episodes of care and not number of actual participants.) | 12 (The enrollment reflects episodes of care and not number of actual participants.)
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Each arm included 12 observations of an episode of care independent of the person being treated. By design of the study, some individuals may have been observed more than once and there may have been fewer than 12 actual participants in each arm.
Groups:
- Trastuzumab Single-Use Injection Device: Participants with HER2-positive EBC received trastuzumab via single-use injection device as 600 mg on Day 1 of each 3-week cycle for a total of 18 cycles. Trastuzumab was supplied in the MO22982 (NCT01401166) trial and dosed according to local labeling.
- Trastuzumab SC Injection: Participants with HER2-positive EBC received trastuzumab via SC injection using vial/syringe as 600 mg on Day 1 of each 3-week cycle for a total of 18 cycles. Trastuzumab was supplied in the MO22982 (NCT01401166) trial and dosed according to local labeling.
- Trastuzumab IV Infusion: Participants with HER2-positive EBC received trastuzumab via IV infusion as 6 mg/kg on Day 1 of each 3-week cycle for a total of 18 cycles. An initial loading dose of 8 mg/kg was given during the first cycle, and also reserved as a reloading dose if treatment was delayed >1 week. Trastuzumab was supplied in the MO22982 (NCT01401166) trial and dosed according to local labeling.
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Single-Use Injection Device | Trastuzumab SC Injection | Trastuzumab IV Infusion | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — The study observed resources required for provision of episodes of care delivered by health care professionals (HCPs). The focus of the observation was the HCP rather than the person being treated, so no demographic data were collected. | NA (NA) — The study observed resources required for provision of episodes of care delivered by HCPs. The focus of the observation was the HCP rather than the person being treated, so no demographic data were collected. | NA (NA) — The study observed resources required for provision of episodes of care delivered by HCPs. The focus of the observation was the HCP rather than the person being treated, so no demographic data were collected. | NA (NA) — The study observed resources required for provision of episodes of care delivered by HCPs. The focus of the observation was the HCP rather than the person being treated, so no demographic data were collected.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — The study observed resources required for provision of episodes of care delivered by HCPs. The focus of the observation was the HCP rather than the person being treated, so no demographic data were collected. | NA — The study observed resources required for provision of episodes of care delivered by HCPs. The focus of the observation was the HCP rather than the person being treated, so no demographic data were collected. | NA — The study observed resources required for provision of episodes of care delivered by HCPs. The focus of the observation was the HCP rather than the person being treated, so no demographic data were collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — The study observed resources required for provision of episodes of care delivered by HCPs. The focus of the observation was the HCP rather than the person being treated, so no demographic data were collected. | NA — The study observed resources required for provision of episodes of care delivered by HCPs. The focus of the observation was the HCP rather than the person being treated, so no demographic data were collected. | NA — The study observed resources required for provision of episodes of care delivered by HCPs. The focus of the observation was the HCP rather than the person being treated, so no demographic data were collected. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Monetary Cost of Health Care Resources Used Per Episode of Care in Administration of Trastuzumab Single-Use Injection Device
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. HCP time was estimated using hourly salary data from National Health Service (NHS) reference costs. Consumable supplies were costed using hospital pharmacy data and online sources. Analysis was limited to only those items with an individual cost of £0.05 or more. Monetary cost of health care resources was determined by adding the costs of consumable supplies and HCP time spent in the administration of trastuzumab single-use injection device during a single episode of care. The average monetary cost per episode was calculated and expressed in pounds.
Time Frame: Data collection up to 1 year
Population: Total Sample: All observations of an episode of care for the given treatment route.
Measure: Mean (Standard Deviation); unit: pounds
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab Single-Use Injection Device
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
pounds | 33.03 (7.69)

2. Primary Outcome: Monetary Cost of Health Care Resources Used Per Episode of Care in Administration of Trastuzumab SC Injection
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. HCP time was estimated using hourly salary data from NHS reference costs. Consumable supplies were costed using hospital pharmacy data and online sources. Analysis was limited to only those items with an individual cost of £0.05 or more. Monetary cost of health care resources was determined by adding the costs of consumable supplies and HCP time spent in the administration of trastuzumab SC injection during a single episode of care. The average monetary cost per episode was calculated and expressed in pounds.
Time Frame: Data collection up to 1 year
Population: Total Sample
Measure: Mean (Standard Deviation); unit: pounds
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab SC Injection
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
pounds | 33.15 (10.74)

3. Secondary Outcome: Monetary Cost of Health Care Resources Used Per Episode of Care in Preparation and Administration of Trastuzumab IV Infusion
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. HCP time was estimated using hourly salary data from NHS reference costs. Consumable supplies were costed using hospital pharmacy data and online sources. Analysis was limited to only those items with an individual cost of £0.05 or more. Monetary cost of health care resources was determined by adding the costs of consumable supplies and HCP time spent in the preparation and administration of trastuzumab IV infusion during a single episode of care. The average monetary cost per episode was calculated and expressed in pounds.
Time Frame: Data collection up to 1 year
Population: Total Sample
Measure: Mean (Standard Deviation); unit: pounds
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab IV Infusion
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
pounds
  Preparation | 22.07 (5.05)
  Administration | 122.89 (14.88)

4. Secondary Outcome: Task-Specific HCP Time Required Per Episode of Care in the Administration of Trastuzumab Single-Use Injection Device
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. HCP time spent on each pre-specified task in the administration of trastuzumab single-use injection device was recorded during each episode of care. The average task-specific HCP time per episode was calculated and expressed in minutes.
Time Frame: Data collection up to 1 year
Population: Total Sample; number (n) of observations per task are shown.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab Single-Use Injection Device
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
minutes
  Pre-infusion set-up (n=9) | 4.0 (2.4)
  Drug collection and check (n=10) | 4.2 (4.0)
  Drug administration (n=12) | 6.1 (0.5)
  Remove and discard device (n=12) | 1.4 (1.1)
  Post-administration monitoring (n=5) | 2.2 (1.1)
  Patient discharge (n=6) | 2.2 (1.9)

5. Secondary Outcome: Task-Specific HCP Time Required Per Episode of Care in the Administration of Trastuzumab SC Injection
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. HCP time spent on each pre-specified task in the administration of trastuzumab SC injection was recorded during each episode of care. The average task-specific HCP time per episode was calculated and expressed in minutes.
Time Frame: Data collection up to 1 year
Population: Total Sample; number (n) of observations per task are shown.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab SC Injection
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
minutes
  Pre-infusion set-up (n=9) | 2.9 (1.8)
  Drug preparation (n=12) | 12.5 (9.1)
  Pre-administration monitoring (n=8) | 3.5 (3.1)
  Drug administration (n=12) | 5.3 (2.2)
  Remove and discard device (n=3) | 0.3 (0.6)
  Post-administration monitoring (n=9) | 1.9 (0.8)
  Patient discharge (n=7) | 1.4 (0.8)

6. Secondary Outcome: Task-Specific HCP Time Required Per Episode of Care in the Administration of Trastuzumab IV Infusion
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. HCP time spent on each pre-specified task in the administration of trastuzumab IV infusion was recorded during each episode of care. The average task-specific HCP time per episode was calculated and expressed in minutes.
Time Frame: Data collection up to 1 year
Population: Total Sample; number (n) of observations per task are shown.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab IV Infusion
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
minutes
  Pre-infusion set-up (n=12) | 8.6 (4.3)
  Drug collection and check (n=9) | 4.6 (3.0)
  Drug administration (n=12) | 32.5 (2.1)
  Monitoring during administration (n=4) | 2.5 (1.9)
  Saline flush (n=12) | 9.4 (6.5)
  Remove and discard supplies (n=11) | 1.6 (0.8)
  Post-administration monitoring (n=2) | 3.0 (1.4)
  Patient discharge (n=9) | 1.8 (1.1)

7. Secondary Outcome: Task-Specific HCP Time Required Per Episode of Care in the Preparation of Trastuzumab IV Infusion
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. HCP time spent on each pre-specified task in the preparation of trastuzumab IV infusion was recorded during each episode of care. The average task-specific HCP time per episode was calculated and expressed in minutes.
Time Frame: Data collection up to 1 year
Population: Total Sample; number (n) of observations per task are shown.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab IV Infusion
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
minutes
  Prepare worksheet (n=9) | 4.6 (3.0)
  Decontamination before aseptic unit (n=12) | 7.2 (5.6)
  Ingredient check (n=12) | 2.3 (1.6)
  Decontamination in aseptic unit (n=11) | 20.7 (15.0)
  Final product check and release (n=12) | 2.6 (1.2)

8. Secondary Outcome: Total HCP Time Required Per Episode of Care in the Administration of Trastuzumab Single-Use Injection Device
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. HCP time spent on each pre-specified task in the administration of trastuzumab single-use injection device was recorded during each episode of care. Total HCP time was determined by adding together the time spent on all tasks. The average total HCP time per episode was calculated and expressed in minutes.
Time Frame: Data collection up to 1 year
Population: Total Sample
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab Single-Use Injection Device
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
minutes | 16.0 (3.9)

9. Secondary Outcome: Total HCP Time Required Per Episode of Care in the Administration of Trastuzumab SC Injection
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. HCP time spent on each pre-specified task in the administration of trastuzumab SC injection was recorded during each episode of care. Total HCP time was determined by adding together the time spent on all tasks. The average total HCP time per episode was calculated and expressed in minutes.
Time Frame: Data collection up to 1 year
Population: Total Sample
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab SC Injection
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
minutes | 24.6 (13.2)

10. Secondary Outcome: Total HCP Time Required Per Episode of Care in the Administration of Trastuzumab IV Infusion
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. HCP time spent on each pre-specified task in the administration of trastuzumab IV infusion was recorded during each episode of care. Total HCP time was determined by adding together the time spent on all tasks. The average total HCP time per episode was calculated and expressed in minutes.
Time Frame: Data collection up to 1 year
Population: Total Sample
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab IV Infusion
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
minutes | 58.1 (5.8)

11. Secondary Outcome: Total HCP Time Required Per Episode of Care in the Preparation of Trastuzumab IV Infusion
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. HCP time spent on each pre-specified task in the preparation of trastuzumab IV infusion was recorded during each episode of care. Total HCP time was determined by adding together the time spent on all tasks. The average total HCP time per episode was calculated and expressed in minutes.
Time Frame: Data collection up to 1 year
Population: Total Sample
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab IV Infusion
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
minutes | 34.5 (13.6)

12. Secondary Outcome: Number of Consumable Medical Supplies Used Per Episode of Care in the Administration of Trastuzumab Single-Use Injection Device
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. Consumable medical supplies used in the administration of trastuzumab single-use injection device were counted during a single episode of care. The average number of each type of consumable used per episode was calculated.
Time Frame: Data collection up to 1 year
Population: Consumables Sample for Trastuzumab Single-Use Injection Device: All observations of an episode of care with trastuzumab single-use injection device that utilized any of the recorded consumable supplies; number (n) of observations per item are shown.
Measure: Mean (Standard Deviation); unit: consumables
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab Single-Use Injection Device
Number analyzed (Participants) | 11
Number analyzed (Episodes of Care) | 11
consumables
  Alcohol swabs (n=11) | 1.2 (0.4)
  Aprons (n=7) | 1.0 (0)
  Dressing packs (n=3) | 1.0 (0)
  Gauze swabs (n=6) | 1.2 (0.4)
  Pairs of gloves (n=10) | 1.6 (0.5)
  Small plasters (n=7) | 1.0 (0)

13. Secondary Outcome: Number of Consumable Medical Supplies Used Per Episode of Care in the Administration of Trastuzumab SC Injection
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. Consumable medical supplies used in the administration of trastuzumab SC injection were counted during a single episode of care. The average number of each type of consumable used per episode was calculated.
Time Frame: Data collection up to 1 year
Population: Consumables Sample for Trastuzumab SC Injection: All observations of an episode of care with trastuzumab SC injection that utilized any of the recorded consumable supplies; number (n) of observations per item are shown.
Measure: Mean (Standard Deviation); unit: consumables
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab SC Injection
Number analyzed (Participants) | 8
Number analyzed (Episodes of Care) | 8
consumables
  Alcohol swabs (n=6) | 1.3 (0.5)
  Aprons (n=6) | 1.0 (0)
  Dressing packs (n=8) | 1.0 (0)
  Gauze swabs (n=4) | 1.0 (0)
  Pairs of gloves (n=7) | 1.6 (0.5)
  Small plasters (n=7) | 1.0 (0)
  10-milliliter (mL) syringes (n=4) | 1.0 (0)
  Mepore dressings (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  Blue needles (n=3) | 1.0 (0)
  Clini-wipes (n=3) | 1.0 (0)
  25-gauge needles (n=2) | 1.0 (0)
  Chloraprep swabs (n=2) | 1.0 (0)
  Wound care packs (n=2) | 1.0 (0)
  Mepore 9x10-centimeter (cm) dressings (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  5-mL syringes (n=6) | 1.0 (0)
  Orange needles (n=7) | 1.0 (0)
  Needles (n=2) | 1.0 (0)
  6-mL syringes (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  Green needles (n=3) | 1.0 (0)
  Leukomed T dressings (n=2) | 1.0 (0)
  Syringes (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  Alco wipes (n=4) | 1.3 (0.5)
  Syringe caps (n=4) | 1 (0)
  20-mL Industrial Molding Supply (IMS) sprays (n=2) | 1 (0)
  10-mL IMS sprays (n=1) | 1 (NA) — Standard deviation not applicable for a single observation (n=1).

14. Secondary Outcome: Number of Consumable Medical Supplies Used Per Episode of Care in the Administration of Trastuzumab IV Infusion
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. Consumable medical supplies used in the administration of trastuzumab IV infusion were counted during a single episode of care. The average number of each type of consumable used per episode was calculated.
Time Frame: Data collection up to 1 year
Population: Consumables Sample for Trastuzumab IV Infusion: All observations of an episode of care with trastuzumab IV infusion that utilized any of the recorded consumable supplies; number (n) of observations per item are shown.
Measure: Mean (Standard Deviation); unit: consumables
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab IV Infusion
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
consumables
  Alcohol swabs (n=12) | 1.5 (0.8)
  Aprons (n=8) | 2.8 (0.7)
  Connectors (n=8) | 1.1 (0.4)
  Dressing packs (n=6) | 1.5 (0.5)
  Gauze swabs (n=7) | 2.3 (1.9)
  Giving sets (n=12) | 1.0 (0)
  Pairs of gloves (n=12) | 3.0 (1.0)
  IV access equipment sets (n=11) | 1.5 (0.9)
  Saline flushes (n=7) | 1.7 (0.8)
  Small plasters (n=11) | 1.1 (0.3)
  10-mL syringes (n=4) | 2.0 (1.2)
  Tegaderm IV dressings (n=10) | 1.3 (0.7)
  100-mL saline (n=9) | 1.6 (0.5)
  Concept wound care packs (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  Tourniquets (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  10-mL heparinised saline (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  50-mL saline (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  21-gauge needles (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  Mepore dressings (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  50-unit heparin (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  Blue needles (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  5-mL heparin (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  250-mL saline (n=1) | 2.0 (NA) — Standard deviation not applicable for a single observation (n=1).

15. Secondary Outcome: Number of Consumable Medical Supplies Used Per Episode of Care in the Preparation of Trastuzumab IV Infusion
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. Consumable medical supplies used in the preparation of trastuzumab IV infusion were counted during a single episode of care. The average number of each type of consumable used per episode was calculated.
Time Frame: Data collection up to 1 year
Population: Consumables Sample for Trastuzumab IV Infusion; number (n) of observations per item are shown.
Measure: Mean (Standard Deviation); unit: consumables
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab IV Infusion
Number analyzed (Participants) | 12
Number analyzed (Episodes of Care) | 12
consumables
  100-mL water injections (n=4) | 1.0 (0)
  10-mL syringes (n=12) | 3.0 (1.7)
  10-mL water injections (n=8) | 4.0 (0.9)
  19-gauge needles (n=6) | 2.7 (2.6)
  21-gauge needles (n=8) | 2.6 (1.8)
  23-gauge needles (n=2) | 3.5 (0.7)
  250-mL saline bags (n=12) | 1.0 (0)
  30-mL syringes (n=3) | 1.0 (0)
  Alco/IMS wipes (n=10) | 5.8 (3.3)
  Pairs of gloves (n=4) | 2.3 (1.3)
  20-mL IMS sprays (n=4) | 1.0 (0)
  50-mL IMS sprays (n=3) | 1.0 (0)
  0.2-cm Minisart filters (n=4) | 1.0 (0)
  Dressing packs (n=2) | 1.0 (0)
  1-mL syringes (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  10-mL sodium chloride (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  Aprons (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  50-mL syringes (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  Infusion hubs (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).
  Baxter caps (n=1) | 1.0 (NA) — Standard deviation not applicable for a single observation (n=1).

16. Secondary Outcome: Total Participant Time Per Episode of Care Spent in the Care Unit for Administration of Trastuzumab
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. Arrival and discharge times were recorded to determine the total time spent in the care unit during a single episode of care. The average time spent in the care unit per episode was calculated and expressed in minutes.
Time Frame: Data collection up to 1 year
Population: Total Sample
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab Single-Use Injection Device | Trastuzumab SC Injection | Trastuzumab IV Infusion
Number analyzed (Participants) | 12 | 12 | 12
Number analyzed (Episodes of Care) | 12 | 12 | 12
minutes | 56.7 (30.3) | 30.3 (14.9) | 94.5 (29.7)

17. Secondary Outcome: Total Participant Time Per Episode of Care Spent in the Chair for Administration of Trastuzumab
Description: The study observed 36 episodes of care (12 per study arm) to collect data on infusion/injection-related tasks. Start and stop 'chair' times were recorded to determine the total time spent in the treatment chair during a single episode of care. The average time spent in the chair per episode was calculated and expressed in minutes.
Time Frame: Data collection up to 1 year
Population: Total Sample
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Episodes of Care
Arm/Group | Trastuzumab Single-Use Injection Device | Trastuzumab SC Injection | Trastuzumab IV Infusion
Number analyzed (Participants) | 12 | 12 | 12
Number analyzed (Episodes of Care) | 12 | 12 | 12
minutes | 30.0 (14.4) | 19.8 (12.4) | 75 (20.9)

ADVERSE EVENTS:
Time Frame: From arrival to discharge during each episode of care (data collection up to 1 year)
Description: Each arm included 12 observations of an episode of care independent of the person being treated. By design of the study, some individuals may have been observed more than once and there may have been fewer than 12 actual participants in each arm.
Arm/Group | Trastuzumab Single-Use Injection Device | Trastuzumab SC Injection | Trastuzumab IV Infusion
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
The focus of the observation in this study was the HCP rather than the person being treated, so number of observations is reported everywhere instead of number of participants. Number of participants was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.